CLINICAL TRIAL: NCT02554058
Title: Phase 1 Effects of Training With a Novel Rehabilitation Bike on the Functional Recovery and Corticospinal Plasticity in Individuals With Incomplete Spinal Cord Injuries
Brief Title: Combined Tactile and Proprioception Training After Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr. Cheryl Glazebrook, Associate Professor, University of Manitoba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Bannatyne2010:157
Record Dates: First submitted 2014-09-05; First posted 2015-09-18 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Spinal Cord Injury
Keywords: Spinal cord injury; rehabilitation; cycling
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cycling and Mechanical stimulation (Experimental): Cycling and Mechanical stimulation : 30 minute cycling training, 3 times a week for 8 weeks.
  Interventions: Device: Cycling and Mechanical stimulation

INTERVENTIONS:
Device: Cycling and Mechanical stimulation — Cycling and Mechanical stimulation : 30 minute cycling training, 3 times a week for 8 weeks.

SUMMARY:
A novel rehabilitation bike has been developed for patients with incomplete spinal cord injuries that incorporates mechanical stimulators on the bike pedals to stimulate the sensory receptors in the soles of the feet; the effect of mechanical stimulator on muscle strengthening has been reported by NASA to improve muscle atrophy in astronauts in zero-gravity environments. Cycling also stimulates lower limb position sensors. We predict that the combination of mechanical stimulation with cycling may be similar enough to walking over ground to lead to gains in balance and mobility. The present study will evaluate the therapeutic effect of this bike on balance, walking, as well as cortical-spinal and spinal pathways in patients with incomplete spinal cord injuries.

DETAILED DESCRIPTION:
INTRODUCTION:

Individuals with spinal cord injuries (SCI) experience balance impairments and limitations in walking. Newer research demonstrates that even after several years individuals with incomplete SCIs can make significant gains in function when they are engaged in targeted physical activity. Previous studies using functional electrical stimulation and locomotion training report reduced spasticity and reflex control, increased electromyography activity during stepping, and increased thigh muscles mass. However, these methods and instruments are bulky, expensive, need technical maintenance, and must be used in a clinical setting. A novel rehabilitation bicycle that uses simultaneous stimulation of plantar mechanoreceptors and hip joint proprioceptors was developed in the department of Biomedical Engineering of University of Manitoba. An advantage of this device is that patients can use it at home and with minimal assistance. Five patients completed initial pilot testing and exhibited an overall improvement on the Berg Balance Scale. Presently, the effect of rehabilitation bike training on the plasticity of the spinal and corticospinal neuronal circuitry and consequently its effects on the functional walking capacity are unclear.

OBJECTIVES:

The purpose of the present study is to evaluate the effect of the rehabilitation bike on corticospinal and spinal plasticity, and functional walking and balance in incomplete SCI individuals.

METHODS:

Ten individuals with chronic incomplete SCI will participate in this study. The protocol will include 30 minute training sessions, three times/week, for 8 weeks. The study design will be a before-after clinical trial with two baseline assessments prior to training. Post-training evaluation after two weeks will be done and there will be a post-training follow-up assessment after two weeks.

Evaluations of functional recovery and independence include: Six -Minute and Ten-Meter Walk Tests, Walking index for spinal cord injury(WISCI II). The Berg Balance Scale(BBS) will be conducted to assess balance. Results will be compared before and after training. H-reflex and motor evoked potential (using transcranial magnetic stimulation ,TMS) will also be measured before and after cycling training to assess the plasticity at the level of the spine and in the corticospinal pathways respectively.

ANTICIPATED RESULTS:

Compared to locomotion training with treadmills and robotic devices, using the rehabilitation bike is affordable and patients are able to use it independently at home, without the help of a physical therapist or a caregiver. Results of this study will clarify the possible positive effect of training with the rehabilitation bike on the corticospinal reorganization as well as training effects on the functional recovery of balance and walking. If the findings from the present study are consistent with the initial pilot data, then it will provide incomplete SCI patients and their therapists with a new option for rehabilitation that is feasible and cost-effective. Considering the relatively high incidence of SCI in Manitoba, the findings from this study will directly improve quality of life for Manitobans and Canadians living with spinal cord injuries.

ELIGIBILITY:
Inclusion Criteria:

* The participant should have experienced a traumatic spinal cord injury
* American Spinal Injury Association (ASIA) class C or D
* Between 18 and 65 years
* At least 12 months post- injury to ensure stability of the patient's neurological condition
* Should be able to walk 10 meters or more with or without assistance (use of braces or walking aids or parallel bars or moderate assistance of one person)
* Should have range of motion in the lower limb joint sufficient to allow the cycling exercise
* Discharged from all rehabilitation.

Exclusion Criteria:

* Impaired mental capacity
* Any medical contradiction to cycling training
* Degenerative spinal disorder
* Significant diagnosed osteoporosis
* Excessive spasticity in the legs as measured by a score of more than 3 on the Modified Ashworth Scale or any spasticity that limits the possibility of cycling exercise or walking
* Obstructive and/or restrictive pulmonary disease
* Severe spinal and Lower Limb deformities
* Decubitus ulcer in the area in contact with the bike and bike's bed

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-05; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in Peak-to-peak amplitude of the motor evoked potentials (MEPs) | 2 weeks prior to first baseline measurement, prior to first training session, after 4 weeks and 8 weeks of training, 2 weeks after the last training session
  MEPs in tibialis anterior muscle using single pulse transcranial magnetic stimulation will be measure.The average of 4 trials in different stimulation intensity will be calculated.
Change in Peak-to-peak amplitude of the H-reflex | 2 weeks prior to first baseline measurement, prior to first training session, after 4 weeks and 8 weeks of training, 2 weeks after the last training session
  Average of 10 peak to peak amplitudes of the H-reflex in soleus muscle with stimulation frequencies of 0.1, 0.2, 0.5 and 10 Hz.

SECONDARY OUTCOMES:
Change in Berg Balance Scale score(BBS) | 2 weeks prior to first baseline measurement, prior to first training session, after 4 weeks and 8 weeks of training, 2 weeks after the last training session
  BBS is a 14-item scale to assess balance.Total Score is 56 points.
Change in 10 meter walk test time | 2 weeks prior to first baseline measurement, prior to first training session, after 4 weeks and 8 weeks of training, 2 weeks after the last training session
  Duration of walking for 10 meters.
Change in 2 minute walk test score | 2 weeks prior to first baseline measurement, prior to first training session, after 4 weeks and 8 weeks of training, 2 weeks after the last training session
  The distance walked within 6 minutes.
Change in Walking index for spinal cord injury (WISCI II) score | 2 weeks prior to first baseline measurement, prior to first training session, after 4 weeks and 8 weeks of training, 2 weeks after the last training session
  WISCI II is an index; it scores the ability of an individual to walk after SCI after a 10 meters of walking. The index score range is 0-20 from the level of most severe impairment (0) to least severe impairment (20) based on the use of devices, braces and physical assistance of one or more persons

OTHER OUTCOMES:
Change in Modified Ashworth Scale score | 2 weeks prior to first baseline measurement, prior to first training session, after 4 weeks and 8 weeks of training
  Modified Ashworth Scale measures muscle tone, or spasticity ( bilateral major hip and knee muscle groups will be assessed clinically in this study).The scores range from 0-4.

CONTACTS AND LOCATIONS:
Overall Officials: Chery Glazebrook, Principal Investigator — University of Manitoba
Locations (1):
- Rehab/Resp Hospital (Health Sciences Center), Winnipeg, Manitoba, Canada